CLINICAL TRIAL: NCT01887938
Title: An Open-Label Extension of Study HGT-MLD-070 Evaluating Long Term Safety and Efficacy of Intrathecal Administration of HGT-1110 in Patients With Metachromatic Leukodystrophy
Brief Title: An Efficacy and Safety Study of HGT-1110 in Participants With Metachromatic Leukodystrophy
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Collaborators: Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HGT-MLD-071; 2012-003775-20 (EudraCT Number); 2024-514403-34-00 (EU CTIS Number)
Record Dates: First submitted 2013-06-20; First posted 2013-06-27 (Estimated); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Metachromatic Leukodystrophy (MLD)
MeSH Terms: conditions — Leukodystrophy, Metachromatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): Participants will receive 10 milligram (mg) of HGT-1110 (Recombinant human arylsulfatase A) intrathecal (IT) injection every-other-week (EOW).
  Interventions: Biological: HGT-1110
- Cohort 2 (Experimental): Participants will receive 30 mg of HGT-1110 IT injection EOW.
  Interventions: Biological: HGT-1110
- Cohort 3 (Experimental): Participants will receive 100 mg of HGT-1110 IT injection EOW.
  Interventions: Biological: HGT-1110
- Cohort 4 (Experimental): Participants will receive 100 mg of HGT-1110 IT injection once weekly for 12 weeks followed by 150 mg EOW.
  Interventions: Biological: HGT-1110

INTERVENTIONS:
Biological: HGT-1110 — Participants will receive IT injection of HGT-1110.
  Other Names: Recombinant human arylsulfatase A

SUMMARY:
The purpose of this study is to collect long-term safety data in participants with metachromatic leukodystrophy (MLD) who are receiving HGT-1110 and have participated in Study HGT-MLD-070 (NCT01510028) through Week 40.

DETAILED DESCRIPTION:
MLD is an inherited, autosomal recessive disorder of lipid metabolism characterized by deficient activity of the lysosomal enzyme, arylsulfatase A (ASA). MLD is a rare orphan disease that occurs in most parts of the world. The estimated overall incidence of the disease in the western world is approximately 1 in 100,000 live births that varies by geographic location. There are no approved therapies for MLD.

This study is a multicenter open-label study designed to evaluate safety and efficacy outcomes of HGT-1110 administered intrathecally in children with MLD who have participated in the dose escalation study, HGT-MLD-070 (NCT01510028), through Week 40 and are receiving study drug every other week (EOW).

Treatment groups will be identical to those in HGT-MLD-070 (NCT01510028), ie, participants assigned to Cohort 1 in Study HGT-MLD-070 (NCT01510028) will continue to receive a dose of 10 milligrams (mg), participants assigned to Cohort 2 in Study HGT-MLD-070 (NCT01510028) will continue to receive a dose of 30 mg, and participants assigned to Cohorts 3 and 4 in Study HGT-MLD-070 (NCT01510028) will continue to receive a dose of 100 mg. Participants in Cohort 4 are to exclusively receive drug product produced with Process B in Study HGT-MLD-070 (NCT01510028) and will continue receiving this drug product in this study. Participants enrolled in this study from Cohorts 1 to 3 in Study HGT-MLD-070 (NCT01510028) were transitioned to Process B after all necessary approvals were obtained. In HGT-MLD-071, all participants in the 10 mg dose cohort who experienced disease progression, as determined by the Investigator, increased to the 30 mg dose after agreement by the Medical Monitor. Based on the interim analysis results from HGT-MLD-070 (NCT01510028 [Cohorts 1-3]), the dose of HGT-1110 will be increased to 100 mg for all participants in HGT-MLD-071 after all necessary approvals were obtained.

ELIGIBILITY:
Inclusion Criteria:

1. Participant has participated in Study HGT-MLD-070 (NCT01510028) through Week 40.
2. Participant must have no safety or medical issues that contraindicate participation.
3. The participant, participant's parent(s), or legally authorized representative(s) must provide written informed consent and/or assent (if applicable) prior to performing any study-related activities.

Exclusion Criteria:

1. The participant is unable to comply with the protocol (example, is unable to return for safety evaluations, or is otherwise unlikely to complete the study) as determined by the investigator.
2. Undergoes bone marrow transplant (BMT), hematopoietic stem cell transplantation (HSCT), or gene therapy at any point during the study.
3. The participant has any known or suspected hypersensitivity to agents used for anesthesia or is thought to be at an unacceptably high risk for associated potential complications of airway compromise or other conditions.
4. The participant is pregnant or breastfeeding.
5. The participant is enrolled in another clinical study that involves clinical investigations or use of any investigational product (drug or drug delivery device) other than those used in HGT-MLD-070 (NCT01510028) within 6 months prior to study enrollment or at any time during the study.
6. The participant has a condition that is contraindicated as described in the SOPH-A-PORT Mini SIDDD Instructions for Use (IFU), including:

   1. The participant has had, or may have, an allergic reaction to the materials of construction of the SOPH-A-PORT Mini S device.
   2. The participant's body size is too small to support the size of the SOPH-A-PORT Mini S Access Port, as judged by the investigator.
   3. The participant has a known or suspected local or general infection.
   4. The participant is at risk of abnormal bleeding due to a medical condition or therapy.
   5. The participant has one or more spinal abnormalities that could complicate safe implantation or fixation.
   6. The participant has a functioning CSF shunt device.
   7. The participant has shown an intolerance to an implanted device.

Ages: 0 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2013-05-23 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events (TEAEs) | Baseline to Follow-up (Week 628)
  An AE is any noxious, pathologic, or unintended change in anatomical, physiologic, or metabolic function as indicated by physical signs, symptoms, or laboratory changes occurring in any phase of a clinical study, whether or not considered investigational drug product-related. TEAEs are defined as all AEs occurring or worsening at or after the first dose of investigational drug product in HGT-MLD-071 or ongoing from HGT-MLD-070 at the time of enrollment into HGT-MLD-071.
Presence of Anti-HGT-1110 Antibodies in Cerebrospinal Fluid (CSF) and Serum | Baseline until end of the study (Week 624)
  The presence of anti-HGT-1110 antibodies in CSF and serum will be assessed.

SECONDARY OUTCOMES:
Change From Baseline in Motor Function as Assessed by Gross Motor Function Measure (GMFM-88) Total Score at Week 624 | Baseline, Week 624
  The GMFM-88 item scores can be used to calculate a domain-specific percent score for each of the 5 GMFM-88 dimensions, which are the following: Lying and rolling; Sitting; Crawling and kneeling; Standing; Walking, running, and jumping. Each of the 88 items is rated on a 4-point scale: 0=does not initiate; 1=initiates; 2=partially completes; and 3=completes. The GMFM-88 total scores range from 0% (no mobility) to a score of 100%, that is (i.e,) the score that can be obtained by an average 5-year-old or older child with normal motor abilities. The domain-specific percent scores are averaged to obtain the total score (percent).
Change From Baseline in the Adaptive Behavior Composite Standard Score Measured by the Vineland Adaptive Behavior Scales, Second Edition (VABS-II) | Baseline, Week 624
  The VABS-II test measures adaptive behaviors, including the ability to cope with environmental changes, to learn new everyday skills, and to demonstrate independence. This test measures the following 4 key domains: communication, daily living skills, socialization, motor skills, and the adaptive behavior composite (a composite of the other 4 domains). The ABC score ranges from 20 to 160 on which higher scores indicate a higher level of adaptive functioning. A positive change value indicates improvement in adaptive functioning.
Change From Baseline in the Domain-Specific Caregiver Observed Metachromatic Leukodystrophy Functioning and Outcomes Reporting Tool (COMFORT) Scores | Baseline, Week 624
  The COMFORT is a questionnaire that will be used to assess health status and the impact of disease on the ability of participants with MLD to carry out activities of daily life. The questionnaire is organized by 8 domains (that is, Personal Care, Positioning, Transfer or Mobility, Eating, Pain and Discomfort During the Day, Sleep, Emotions, Communication, Play and Leisure Activities) and will be completed by the participant's parent(s) or legal representative(s). It will be conducted in available validated languages. The COMFORT scores range from 0 to 100, with higher scores indicating a decline in the functioning.
Maximum Observed Serum Concentration (Cmax) of HGT-1110 | Pre-dose, 0.5, 1, 2, 4, 8, 12, 24, and 48 hours post-dose on Weeks 104, 258, 364 and 622 in Cohort 4 and Week 8 in Cohorts 1-3
  The Cmax of HGT-1110 will be assessed.
Time of Maximum Observed Serum Concentration (Tmax) of HGT-1110 | Pre-dose, 0.5, 1, 2, 4, 8, 12, 24, and 48 hours post-dose on Weeks 104, 258, 364 and 622 in Cohort 4 and Week 8 in Cohorts 1-3
  The Tmax of HGT-1110 will be assessed.
Area Under the Serum Concentration-Time Curve From Time Zero to the Last Sampling Time at Which Serum Concentrations Were Measurable (AUC0-last) of HGT-1110 | Pre-dose, 0.5, 1, 2, 4, 8, 12, 24, and 48 hours post-dose on Weeks 104, 258, 364 and 622 in Cohort 4 and Week 8 in Cohorts 1-3
  The AUC0-last of HGT-1110 will be assessed.
Area Under the Serum Concentration-Time Curve Extrapolated to Infinity (AUC0-inf) of HGT-1110 | Pre-dose, 0.5, 1, 2, 4, 8, 12, 24, and 48 hours post-dose on Weeks 104, 258, 364 and 622 in Cohort 4 and Week 8 in Cohorts 1-3
  The AUC0-inf of HGT-1110 will be assessed.
Apparent Terminal Rate Constant (lambda z) of HGT-1110 | Pre-dose, 0.5, 1, 2, 4, 8, 12, 24, and 48 hours post-dose on Weeks 104, 258, 364 and 622 in Cohort 4 and Week 8 in Cohorts 1-3
  The lambda z of HGT-1110 will be assessed.
Terminal Half-Life (t1/2) of HGT-1110 | Pre-dose, 0.5, 1, 2, 4, 8, 12, 24, and 48 hours post-dose on Weeks 104, 258, 364 and 622 in Cohort 4 and Week 8 in Cohorts 1-3
  The t1/2 of HGT-1110 will be assessed.
Clearance (CL/F) of HGT-1110 | Pre-dose, 0.5, 1, 2, 4, 8, 12, 24, and 48 hours post-dose on Weeks 104, 258, 364 and 622 in Cohort 4 and Week 8 in Cohorts 1-3
  The CL/F of HGT-1110 will be assessed.
Volume of Distribution (Vz/F) of HGT-1110 | Pre-dose, 0.5, 1, 2, 4, 8, 12, 24, and 48 hours post-dose on Weeks 104, 258, 364 and 622 in Cohort 4 and Week 8 in Cohorts 1-3
  The Vz/F of HGT-1110 will be assessed.
Concentrations of HGT-1110 in Cerebrospinal Fluid (CSF) | Baseline to End of the study (Week 624)
  Concentrations of HGT-1110 in CSF will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (15):
- The Children's Hospital at Westmead, Westmead, Australia
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Brazil
- Detska Interni Klinika, Lf Mu A Fn Brno, Brno, Czechia
- Rigshospitalet, Copenhagen, Denmark
- France (5):
  - Hopital Femme Mere Enfant, Bron
  - Hopital Gui de Chauliac - CHRU de Montpellier, Montpellier
  - CHU de Nantes, Nantes
  - CHR Orleans - Hopital La Source, Orléans
  - Hôpital de Bicêtre, Le Kremlin-Bicêtre, Île-de-France Region
- Germany (3):
  - Center for Pediatric Clinical Studies (CPCS), Tübingen, Baden-Wurttemberg
  - Klinikum Oldenburg, Oldenburg
  - Marien-Hospital Wesel gGmbh, Wesel
- Japan (3):
  - Kitakyushu Municipal Yahata Hospital, Fukuoka
  - Kurashiki Central Hospital, Okayama Prefecture
  - Osaka University Hospital, Osaka

IPD SHARING:
Plan to Share IPD: No
- De-identified individual participant data from this particular study will not be shared as there is a reasonable likelihood that individual patients could be re-identified (due to the limited number of study participants/study sites, …)

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language, including a Plain Language Summary of the results if the trial has been completed. — https://clinicaltrials.takeda.com/study-detail/5f6b5fce4db2bf003ab467a0